CLINICAL TRIAL: NCT06767059
Title: The Effect of Walking and Grounding on Pain Intensity, Fatigue Level, and Sleep Quality in Women With Breast Cancer
Brief Title: The Effect of Walking and Grounding in Women With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Baise Bicav, Science Specialist Lecturer, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AÜ-HEM-BB-01
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Walking; Grounding; Nursing
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Three groups with walking, grounding and control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be told which group they are in the study. To prevent selection bias in the study, the determination of the groups will be made by the nurse outside the study. To prevent omission and reporting bias in the study, the data will be coded with the letters A, B and C without specifying which group they are in. The data will be computerized by a person outside the study. Data will be analyzed coded in terms of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Walking Group (Experimental): Patients will walk for 30 minutes at least 3 times a week.
  Interventions: Other: Walking Group
- Grounding Group (Experimental): Patients will walk with a grounding stick for 30 minutes at least 3 times a week.
  Interventions: Other: Grounding Group
- Control Group (No Intervention): Routine follow-up will be done.

INTERVENTIONS:
Other: Walking Group — Patients will be asked to walk for 30 minutes at least 3 times for 8 weeks. In order to ensure regular follow-up, patients will be asked to write on the walking tracking form when they walk and the number of steps before they start walking and the number of steps after walking using the application.
  Arms: Walking Group
Other: Grounding Group — Patients will be asked to walk with a grounding stick for 30 minutes at least 3 times for 8 weeks. Patients will be asked to fill in the walking follow-up form and grounding follow-up form for regular follow-up.
  Arms: Grounding Group

SUMMARY:
This randomized controlled trial was conducted to examine the effect of walking and grounding on pain intensity, fatigue level and sleep quality in women diagnosed with breast cancer.

DETAILED DESCRIPTION:
Grounding is the flow of electrons by direct contact of the body's natural electric charge with the earth. There are many methods of grounding. Earthing systems can be used while sitting or sleeping, or the cheapest and easiest way is to walk barefoot in a grassy park, garden or beach. Earthing improves circulation by increasing blood flow and oxygenation of each organ system, positively affecting cardiovascular function. Hormones normalize, cortisol drops, blood sugar stabilizes, sleep improves, energy increases and inflammation decreases. When electrical contact between the body and the earth is re-established through grounding, organ system function begins to optimize again. When people are grounded, they feel more alive, healthy and energized than when they are ungrounded. The literature reports that human grounding has many positive effects on pain, sleep and fatigue. Grounding can be an effective method in managing pain, fatigue and sleep problems, which are among the most common problems in patients with breast cancer. Earthing is one of the biggest challenges of the modern world. City life, contact with the land The decline of the earth's energy supply, living and working indoors, and wearing plastic shoes disrupt our natural energy circuit. Although barefoot walking is the cheapest and easiest way to become grounded, dirty soil, foot This method may be a disadvantage for women with breast cancer due to conditions such as wounding of the base. In this study, a conductive device is used for grounding cancer patients by providing indirect contact with the soil.

grounding will be ensured while walking with the stick. While grounding has many positive effects on health, no grounding study was found in the literature review in the field of nursing. This study is a part of both the It is thought to positively affect the pain, fatigue and sleep problems of women with breast cancer by walking with shoes and providing grounding in order to use the positive effects of grounding.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Can read and write and speak Turkish,
* Diagnosed with primary breast cancer and know the diagnosis,
* Volunteered to participate in the research,
* Living in Ankara province,
* Paclitaxel or Paclitaxel-Transtuzumab based chemotherapy treatment initiated,
* Eastern Cooperative Oncology Group (ECOG) Scale 0 or 1,
* NCI-CTCAE v5.0 Pain, fatigue and sleep toxicity grade 1 or 2,
* You have a phone with an iOS or Android processor,

Exclusion Criteria:

* Open wounds or edema of the hands and feet,
* NCI-CTCAE v5.0 motor and sensory peripheral neuropathy with toxicity grade 3,4 or 5,
* People with a disability that would prevent them from walking,
* Diagnosed cardiovascular and pulmonary disorders,
* Diagnosed psychiatric illness,
* Communication problems,
* Bone metastases,
* Bilateral mastectomies,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer is diagnosed more frequently in women.
Enrollment: 54 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 0,4,8 weeks
  It will be used in the study to measure pain, fatigue, and sleep severity. The VAS consists of a measured horizontal or vertical line with definitions such as "no symptoms" or "severe symptoms" at both ends. The severity of the patient's symptoms is measured by marking a numbered point on this line. For pain symptoms, the severity is marked on a 10 cm (100 mm) ruler with "no pain" at one end and "unbearable pain" at the other. The intervals for pain severity are defined as follows: <3 mild pain, 3-6 moderate pain, >6 severe pain. The VAS is a reliable and valid method for assessing pain intensity (Arslan et al., 2016). The VAS will also be used to assess fatigue and sleep intensity. It is marked as 0 none to 10 very much.
  It is measured as 0 none, 1-3 mild, 4-6 moderate, and 7-9 severe.

SECONDARY OUTCOMES:
Visual Similarity Scale for Fatigue | 0,4,8 weeks
  The scale consists of 18 items and two subscales: fatigue (items 1-5, 11-18) and energy (items 6-10). There are 10 cm long horizontal lines with positive and negative statements at one end and negative statements at the other end of the FLSS, respectively. While the items of the fatigue subscale progress from positive to negative, the energy subscale has the opposite order. The lowest score obtained from the fatigue subscale is 0 and the highest score is 130. In the energy subscale, the scores are in the range of 0 to 50. A high score on the fatigue subscale and a low score on the energy subscale indicates that the severity of fatigue is high. In the validity and reliability study of the scale, it was reported that the Cronbach's α internal consistency coefficient for the 13-item fatigue subscale was 0.90 and 0.74 for the 5-item energy subscale.
Pittssburgh Sleep Quality Index | 0,4,8 weeks
  The Pittsburgh sleep quality index is a reliable and consistent sleep questionnaire that includes 24 questions to assess sleep quality, amount of sleep, presence and severity of sleep disturbance in the last one month. Its diagnostic sensitivity is 89.6% and specificity is 86.5%. The PSQI consists of seven components assessing subjective sleep quality, sleep latency, sleep duration, sleep efficiency-established sleep efficiency, sleep disturbance, sleep medication use, and impairment in daytime activities. Some of these components consist of a single question, while others are a grouping of several questions. Scoring consists of the scores given to the questions or groups of questions covered by these components. The sum of the scores of the seven components gives the total PDQI score. Each question is evaluated on a 0-3 point scale. The total score has a value between 0-21. A high total score indicates poor sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Baise Bicav, MSc, Principal Investigator — Ankara University; Sevinç Kutlutürkan, PhD, Principal Investigator — Ankara University
Locations (1):
- Gazi University Health Research and Application Center Gazi Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No